CLINICAL TRIAL: NCT01416038
Title: Phase 1-2 Study of an Immunotherapeutic Vaccine, DPX-Survivac With Low Dose Cyclophosphamide in Patients With Surgically Operable or Advanced Stage Ovarian, Fallopian Tube or Peritoneal Cancer
Brief Title: Phase 1 Study of a Cancer Vaccine to Treat Patients With Advanced Stage Ovarian, Fallopian or Peritoneal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ImmunoVaccine Technologies, Inc. (IMV Inc.) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONC-DPX-Survivac-01
Record Dates: First submitted 2011-08-09; First posted 2011-08-12 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer
Keywords: vaccine; immunotherapy; ovarian; fallopian tube; peritoneal; cancer; tumor; Phase 1; Phase I; combination therapy
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Neoplasms | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Vaccine (Experimental): Cohort A: 0.5 mL of DPX-Survivac (injection)
  Interventions: Biological: DPX-Survivac
- Vaccine + low dose cyclophosphamide (Experimental): Cohort B: 0.1 mL DPX-Survivac (injection) with low dose cyclophosphamide (oral)
  Interventions: Biological: DPX-Survivac; Drug: low dose cyclophosphamide (oral)
- Vaccine + low dose cyclophosphamide. (Experimental): Cohort C: 0.5 mL DPX-Survivac (injection) with low dose cyclophosphamide (oral)
  Interventions: Biological: DPX-Survivac; Drug: low dose cyclophosphamide (oral)

INTERVENTIONS:
Biological: DPX-Survivac — Vaccine targeting survivin antigen will be administered subcutaneously.
Drug: low dose cyclophosphamide (oral) — Low dose cyclophosphamide will be taken by mouth.
  Arms: Vaccine + low dose cyclophosphamide; Vaccine + low dose cyclophosphamide.

SUMMARY:
Immunotherapy is a novel way to treat cancer and does so by targeting the immune system to destroy tumor cells. Many different therapeutic vaccines have been evaluated in phase 1, 2, and even phase 3 trials. Much has been learned about the principles of applying immune-based therapies and specifically the types of patients that may be most likely to mount an effective immune response. When used alone, cancer vaccines may have their greatest impact earlier in the disease course or in situations with minimal residual disease.

ImmunoVaccine Technologies Inc. (Immunovaccine) is an immuno-oncology company developing a novel adjuvanting technology platform termed DepoVax. DepoVax was created to enhance the speed, strength and duration of an immune response. The peptide antigens included in DPX-Survivac are designed to target Survivin, a protein which is over-expressed in many cancer types, including epithelial ovarian cancers.

This study was designed be a phase 1-2 trial to determine the safety and immunogenicity profiles of DPX-Survivac, a therapeutic vaccine co-administered with a regimen of low dose oral cyclophosphamide. The dosing-finding phase 1 study of 15 subjects would move directly into a randomized phase 2 study. However, with the evolving field of immunotherapy Immunovaccine has begun to focus on combination therapies, combining DPX-Survivac treatment with checkpoint inhibitors and other immune modulators, such as in NCT02785250.

DETAILED DESCRIPTION:
The standard treatment for all ovarian cancer is aggressive debulking surgery followed by chemotherapy. Ovarian carcinoma is one of the most chemosensitive solid tumors and early stage patients are most responsive to treatment. However, despite improvements to the standard treatment over the past three decades, almost all patients with advanced stage disease at presentation will relapse, with an average progression free survival of 16-18 months. When residual or recurrent disease manifests itself, resistance to chemotherapy often prohibits further curative therapy. Therefore, there are still significant unmet needs in treating ovarian cancer patients.

Treatment with DPX-Survivac is for patients with late-stage ovarian, fallopian tube, or peritoneal cancer who have completed initial chemotherapy treatment and successful debulking surgery. The phase 1 dose finding study will administer 3 doses of DPX-Survivac with or without accompanying low dose oral cyclophosphamide.

ELIGIBILITY:
Main Inclusion Criteria:

* Subjects with stage IIc-IV epithelial ovarian, fallopian tube and peritoneal cancer who have completed adjuvant treatment consisting of up to 8 cycles of paclitaxel and carboplatin chemotherapy or other acceptable chemotherapy after initial debulking surgery with evidence of a complete or partial response by radiological imaging. These subjects may remain on hormonal therapy during the trial if such treatment has been prescribed by their treating physician. These subjects may have been in a clinical trial for an investigational carboplatin based adjuvant therapy.
* Subjects with recurrent ovarian, fallopian tube or peritoneal cancer who have clinical or radiologic evidence of a complete or partial response or stable disease after completion of first-line chemotherapy for their recurrent disease and are not suitable for additional cytotoxic therapy are eligible. These subjects may have previously received a course of adjuvant chemotherapy earlier in their disease management as described in point one above. These subjects are eligible regardless of their CA-125 results. These subjects may have been in a clinical trial of an investigational therapy.
* Subjects may have received previous courses of an investigational biologic therapy including active or passive immunotherapy greater than 60 days prior to receiving the first injection of DPX-Survivac
* At least 30 days since localized surgery, radiotherapy or chemotherapy
* Subjects may be on a biphosphonate provided it had not been initiated within 14 days prior to receiving the first injection of DPX-Survivac

Main Exclusion Criteria:

* Subjects undergoing concurrent chemotherapy, radiation therapy, immunotherapy are excluded
* Subjects who participated in therapeutic adjuvant ovarian cancer studies are excluded except for platinum-based adjuvant studies
* Subjects who have received more than one course of chemotherapy for recurrent disease
* Subjects receiving bevacizumab for maintenance therapy are excluded (subjects who received bevacizumab as part of their adjuvant therapy will be permitted)
* History of autoimmune disease
* Subjects with recent history of thyroiditis
* Presence of an acute infection requiring antibiotics within 4 weeks of study entry or a chronic infection including but not limited to: urinary tract infection, HIV, viral hepatitis
* Subjects with brain metastases
* Concurrent (within the last 5 years) second malignancy other than non melanoma skin cancer, cervical carcinoma in situ, or controlled bladder cancer
* Acute or chronic skin disorders that will interfere with subcutaneous injection of the vaccine or subsequent assessment of potential skin reactions
* Serious intercurrent chronic or acute illness, such as cardiac disease, hepatic disease, or other illness considered by the investigator as an unwarranted high risk for an investigational product
* Subjects on steroid therapy or other immunosuppressive, such as azathioprine or cyclosporin A
* Allergies to any component of the vaccine
* Pregnant or nursing mothers
* Subjects with a medical or psychological impediment to probable compliance with the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Number of reported adverse events | Until 6 month follow up
  The number of adverse events along with the results of vital sign measurements, physical examinations, and clinical laboratory tests will be used to determine the safety profile of subcutaneous administration of DPX-Survivac.

SECONDARY OUTCOMES:
Levels of cell mediated immunity targeting the survivin epitopes | Until 6 month follow up

CONTACTS AND LOCATIONS:
Locations (7):
- United States (5):
  - Roswell Park Cancer Institute, Buffalo, New York
  - Winthrop University Hospital, Mineola, New York
  - Duke University Medical Center, Durham, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - Mary Crowley Cancer Research Center, Dallas, Texas
- Canada (2):
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Princess Margaret Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Berinstein NL, Karkada M, Oza AM, Odunsi K, Villella JA, Nemunaitis JJ, Morse MA, Pejovic T, Bentley J, Buyse M, Nigam R, Weir GM, MacDonald LD, Quinton T, Rajagopalan R, Sharp K, Penwell A, Sammatur L, Burzykowski T, Stanford MM, Mansour M. Survivin-targeted immunotherapy drives robust polyfunctional T cell generation and differentiation in advanced ovarian cancer patients. Oncoimmunology. 2015 May 7;4(8):e1026529. doi: 10.1080/2162402X.2015.1026529. eCollection 2015 Aug. PMID 26405584